CLINICAL TRIAL: NCT00264316
Title: A Double-blind, Randomised, Controlled Study of Autologous Bone Marrow-Derived Stem Cell Transfer In Patients With ST-Segment Elevation Myocardial Infarction.
Brief Title: Bone Marrow-Derived Stem Cell Transfer in Acute Myocardial Infarctions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: SJ-CAR-ML2170
Record Dates: First submitted 2005-12-09; First posted 2005-12-12 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2005-12

CONDITIONS: Myocardial Infarction
Keywords: bone marrow cell transfer; acute myocardial infarction; left ventricular function
MeSH Terms: conditions — Myocardial Infarction

INTERVENTIONS:
Procedure: bone marrow-derived stem cell transfer

SUMMARY:
The benefit of reperfusion therapies for ST-elevation acute myocardial infarction (STEMI) is limited by postinfarction left ventricular (LV) dysfunction.The purpose of this study is to determine whether intracoronary transfer of bone marrow cells will augment left ventricular function recovery of the heart.

DETAILED DESCRIPTION:
Despite early coronary reperfusion, salvage of ischemic myocardium is incomplete and loss of viable myocardium initiates a process of adverse left ventricular (LV) remodeling1, compromising clinical outcome.

Experimental data have suggested that autologous bone marrow-derived or circulating progenitor cells may be beneficial for LV function recovery, but underlying mechanisms are unclear and prominent cardiomyocyte transdifferentiation has only been reported under selected experimental conditions. Early non-randomized clinical investigations indicate feasibility, safety and enhanced functional recovery after autologous human bone marrow-derived stem cell (BMSC) infusion into the infarct-related artery. More recently, a randomized open study demonstrated improvement of LV systolic function but not of LV remodeling following BMSC transfer.

In the absence of trials, in which the control group reproduces the exact conditions of the cell transfer group, including bone marrow aspiration and a placebo intracoronary injection, the true benefit of cell transfer cannot be fully appreciated.

We, therefore, designed a randomized, double-blind, and placebo-controlled exploratory study to investigate the effect of autologous BMSC transfer on LV functional and structural recovery after myocardial infarction. In view of the exploratory nature of the study and to detect potential mechanisms for the biological effect, we also assessed myocardial perfusion and oxidative metabolism using serial 1-[11C]acetate positron emission tomography (PET).

ELIGIBILITY:
Inclusion Criteria:

* patients with acute myocardial infarction with cumulative ST-segment elevation >=6mm, successful epicardial reperfusion after PCI and significant LV dysfunction

Exclusion Criteria:

* patients presenting within 2 hours of symptom onset (no dilution of any treatment effect from aborted infarctions)
* patients with prior coronary artery bypass grafting, pulmonary edema, cardiogenic shock or significant co-morbidities

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68
Dates: Start 2003-05; Study Completion 2005-12

PRIMARY OUTCOMES:
increase in global LV ejection fraction fraction; evaluation by magnetic resonance (MRI) after 4 months

SECONDARY OUTCOMES:
change in infarct size and regional LV function; evaluation by magnetic resonance (MRI) after 4 months
change in myocardial perfusion and oxidative metabolism; investigated using serial 1-[11C]acetate positron emission tomography after 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Janssens, MD, PhD, Principal Investigator — Department of Cardiology, University Hospital Gasthuisberg, Leuven, Belgium; Frans Van de Werf, MD, PhD, Study Director — Department of Cardiology, University Hospital Gasthuisberg, Leuven, Belgium
Locations (1):
- Department of Cardiology, University Hospital Gasthuisberg, Leuven, Belgium

REFERENCES:
- [Result] Janssens S, Dubois C, Bogaert J, Theunissen K, Deroose C, Desmet W, Kalantzi M, Herbots L, Sinnaeve P, Dens J, Maertens J, Rademakers F, Dymarkowski S, Gheysens O, Van Cleemput J, Bormans G, Nuyts J, Belmans A, Mortelmans L, Boogaerts M, Van de Werf F. Autologous bone marrow-derived stem-cell transfer in patients with ST-segment elevation myocardial infarction: double-blind, randomised controlled trial. Lancet. 2006 Jan 14;367(9505):113-21. doi: 10.1016/S0140-6736(05)67861-0. PMID 16413875